CLINICAL TRIAL: NCT04927936
Title: A Multicenter, Randomised, Single-blind, Controlled Trial Among HealthCare Workers (HCW) Vaccinated With Janssen Vaccine: the SWITCH Trial
Brief Title: A Trial Among HealthCare Workers (HCW) Vaccinated With Janssen Vaccine: the SWITCH Trial
Acronym: SWITCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Leiden University Medical Center (Other); University Medical Center Groningen (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Hugo van der Kuy, Prof dr, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MEC-2021-0132; 2021-000701-24 (EudraCT Number)
Record Dates: First submitted 2021-06-06; First posted 2021-06-16 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: vaccination; heterologous boosting
MeSH Terms: conditions — COVID-19 | interventions — Vaccination

STUDY DESIGN:
Intervention Model Description: A multicenter, randomised, single-blind, controlled trial to determine reactogenicity and immunogenicity of different prime-boost COVID-19 vaccine schedules.
  Setting Multicenter study conducted through 4 academic trial sites (Amsterdam UMC, Erasmus MC, Leiden UMC, and UMC Groningen).
  Trial duration Total duration of each participant will be 12 months from the administration of the boost vaccine dose.
Who Masked: Participant
Masking Description: Participants will be randomised per cohort in 1:1:1:1 fashion using block randomisation.
  The study will be single-blind. Staff involved in study will be aware of which vaccine the participant is receiving (arm allocation); the participants will remain blinded to their vaccine allocation.
  Seven days (after filling in the questionnaires regarding side-effects) after the boost (2nd vaccination) the vaccination strategy will be unblinded. Directly after the boost (2nd vaccination) a letter will be given in which the study is explained and a statement is given that a second vaccination is given.
  Those participants receiving only one shot with Janssen will only be told on the day of planned boost (2nd vaccination). They will not be vaccinated with placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Janssen vaccine only (Active Comparator): HCW already vaccinated with Janssen vaccine once. 84 days after the first vaccination, blood samples will be drawn (day =0, baseline) This will be repeated at day 28 (primary endpoint), day 180 and day 365. This arm will have 87 +25% seropositive for SARS-CoV-2 IgG at baseline or loss to follow-up = 108 participants.
  In this arm half of the participants will undergo a detailed immunological assessment (n=54 per arm).
  Interventions: Biological: Vaccination once with Janssen vaccine (only priming)
- Janssen vaccine - Janssen vaccine (Experimental): HCW already vaccinated with Janssen vaccine once. 84 days after the first vaccination a boost will be given with Janssen vaccine and blood samples will be drawn (day =0, baseline) This will be repeated at day 28 (primary endpoint), day 180 and day 365. This arm will have 87 +25% seropositive for SARS-CoV-2 IgG at baseline or loss to follow-up = 108 participants.
  In this arm half of the participants will undergo a detailed immunological assessment (n=54 per arm).
  Interventions: Biological: Vaccination with Janssen vaccine followed with Janssen vaccine (homologous boosting).
- Janssen vaccine - Moderna vaccine (Experimental): HCW already vaccinated with Janssen vaccine once. 84 days after the first vaccination a boost will be given with Moderna vaccine and blood samples will be drawn (day =0, baseline) This will be repeated at day 28 (primary endpoint), day 180 and day 365. This arm will have 87 +25% seropositive for SARS-CoV-2 IgG at baseline or loss to follow-up = 108 participants.
  In this arm half of the participants will undergo a detailed immunological assessment (n=54 per arm).
  Interventions: Biological: Vaccination with Janssen vaccine followed with Moderna vaccine (heterologous boosting).
- Janssen vaccine - Pfizer vaccine (Experimental): HCW already vaccinated with Janssen vaccine once. 84 days after the first vaccination a boost will be given with Pfizer vaccine and blood samples will be drawn (day =0, baseline) This will be repeated at day 28 (primary endpoint), day 180 and day 365. This arm will have 87 +25% seropositive for SARS-CoV-2 IgG at baseline or loss to follow-up = 108 participants.
  In this arm half of the participants will undergo a detailed immunological assessment (n=54 per arm).
  Interventions: Biological: Vaccination with Janssen vaccine followed with Pfizer vaccine (heterologous boosting).

INTERVENTIONS:
Biological: Vaccination once with Janssen vaccine (only priming) — Vaccination (priming) with janssen vaccine. There is no boosting.
  Arms: Janssen vaccine only
Biological: Vaccination with Janssen vaccine followed with Janssen vaccine (homologous boosting). — Vaccination (priming) with janssen vaccine. There is boosting with Janssen vaccine.
  Arms: Janssen vaccine - Janssen vaccine
Biological: Vaccination with Janssen vaccine followed with Moderna vaccine (heterologous boosting). — Vaccination (priming) with janssen vaccine. There is boosting with Moderna vaccine.
  Arms: Janssen vaccine - Moderna vaccine
Biological: Vaccination with Janssen vaccine followed with Pfizer vaccine (heterologous boosting). — Vaccination (priming) with janssen vaccine. There is boosting with Pfizer vaccine.
  Arms: Janssen vaccine - Pfizer vaccine

SUMMARY:
The key objective of the study is to measure the immune response against SARS-CoV-2 after different vaccinations in Health Care Workers (HCW) from 18 to 65 years old vaccinated once with Janssen vaccine.

Determination of antibodies by a quantitative immunoglobulin G (IgG) assay (LIAISON SARS-CoV-2 TRIMERICS IgG essay) 28 days after second vaccination (booster) comparing, per protocol, the following three groups:

1. Janssen vaccine/- vs. Janssen vaccine/Janssen vaccine
2. Janssen vaccine/Janssen vaccine vs. Janssen vaccine/Pfizer vaccine
3. Janssen vaccine/Janssen vaccine vs. Janssen vaccine/Moderna vaccine

DETAILED DESCRIPTION:
Rationale: A novel coronavirus (SARS CoV-2) was first detected in Wuhan, China in December 2019 (1). In January 2021 the first vaccines protecting against this virus are available in the Netherlands. Most current available vaccines in the Netherlands (e.g., AstraZeneca vaccine (2), Moderna vaccine (3), and Pfizer vaccine (4) require a second boost (2nd vaccination) after the prime (1st vaccination), to obtain an optimal immune response. The booster (2nd vaccination) has up to present always been given with the same vaccine as the primary vaccine. Unfortunately, the availability of the vaccines is limited and a speedy vaccination is also hampered by logistic reasons. The ability to combine different vaccines could make vaccination programs in the future more flexible. It would facilitate a fast-track process and reduce the impact of any supply-chain disruptions (5). In addition, several studies in mice have already shown that combining different vaccines (two-dose heterologous vaccination regimen) can elicit a broader immune response (in field of neutralizing antibodies and T-cell responses)(6, 7). These results endorse the need for clinical trials to investigate the immunogenicity of heterologous regimens. Trails to combine different vaccines have meanwhile been set up in Great Britain and Spain where they combine Pfizer vaccine and AstraZeneca vaccine (Com-COV 1(8) and CombiVacS(9)). Recently, it became known that the CoM-COV1 was expanded with Moderna vaccine and Novavax vaccine (CoM-COV2(10)). Therefore this protocol has a focus to adeno priming with Janssen vaccine, which is not studied in the other ongoing studies. As the vaccination rate in The Netherlands is increasing rapidly, it was decided to include Healthcare Workers (HCW) vaccinated once with Janssen vaccine. Objective: The key objective of the study is to measure the immune response against SARS-CoV-2 after different vaccinations in Health Care Workers (HCW) from 18 to 65 years old.

Determination of antibodies by a quantitative IgG assay (LIAISON SARS-CoV-2 TrimericS IgG essay) 28 days after second vaccination (booster) comparing, per protocol, the following three groups:

1. Janssen vaccine/- vs. Janssen vaccine/Janssen vaccine
2. Janssen vaccine/Janssen vaccine vs. Janssen vaccine/Pfizer vaccine
3. Janssen vaccine/Janssen vaccine vs. Janssen vaccine/Moderna vaccine Study design: A multicenter, randomised, single-blind, controlled trial to determine reactogenicity and immunogenicity of different prime-boost COVID-19 vaccine schedules.

Setting: multicenter study conducted at 4 academic University Medical Centers (UMC) hospitals (Amsterdam UMC, Erasmus UMC, Leiden UMC, and UMC Groningen).

Hypothesis: Immunogenicity in participants who have already received one dose of Janssen vaccine will be higher when it is followed by a heterologous booster containing Pfizer vaccine or Moderna vaccine as opposed to a homologous booster containing Janssen vaccine.

The main question that will be addressed: Measuring the humoral immune response against SARS-CoV-2 after inoculation with a single-dose Janssen vaccine compared to a homologous vaccination regimen with Janssen vaccine/Janssen vaccine and the comparison of a homologous vaccination regimen (Janssen vaccine/Janssen vaccine) with a heterologous vaccination regimen (Janssen vaccine/Pfizer vaccine + Janssen vaccine/Moderna vaccine).

Participants will be randomized for Standard of Care (1 vaccination with Janssen vaccine), a homologue vaccination strategy (two vaccines from the same manufacturer, i.e., Janssen vaccine) or a heterologous vaccination strategy (two different vaccines, e.g., Janssen vaccine followed by Pfizer vaccine or Moderna vaccine). The study starts approximately 84 days (+/- 10) after the first vaccination Janssen vaccine. The day of the 2nd vaccination is seen as day 0. Blood will be drawn at 4 different time points, i.e. day 0 - baseline (before 2nd vaccination), day 28 (after 2nd vaccination - primary endpoint), day 180 +/- 14 days (after 2nd vaccination), and day 365 +/- 14 days (after 2nd vaccination). Questionnaires will be used to monitor for adverse reactions after 2nd vaccination and to evaluate COVID-19 infection during the study and outcome despite vaccination.

Study population: Healthcare Workers (HCW) from 18 to 65 years old vaccinated once with Janssen vaccine. Individuals of all ethnicities will be recruited. Given the speed of the Dutch vaccination campaign, it is not feasible to collect baseline immunological data before first vaccination. For this reason, the baseline in this study is at the day of the booster (2nd vaccination). If not enough HCW can be found within the recruiting hospitals, the population will be expanded to HCW in surrounding peripheral hospitals and primary care (e.g., local pharmacies, dental practices, and physiotherapists).

Intervention (if applicable): All adult people in the Dutch population are vaccinated on a voluntary basis. The only difference is that they might be vaccinated with a different vaccine for the boost (second vaccination).

Main study parameters/endpoints:

Primary endpoint: to determine whether the immune response 28 days after boost is higher to that observed following only one vaccination (Janssen vaccine solo vs. Janssen vaccine/Janssen vaccine) and the comparison of a heterologous boost of a COVID-19 vaccine (84 days post prime (1st vaccination) - Janssen vaccine/Pfizer vaccine and Janssen vaccine/Moderna vaccine) with a homologous boost (84 days post prime (1st vaccination) - Janssen vaccine/Janssen vaccine), in participants vaccinated once with Janssen vaccine.

Secondary endpoints: to assess safety & reactogenicity of different prime-boost schedules of COVID-19 vaccines and characterization of immunogenicity of different prime-boost schedules of COVID-19 vaccines.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The consequence of participating in this study has two sides; on the one hand, a higher burden for the participant, given 4 study visits in one year including blood samples and questionnaires. With the fact that slightly more side effects may be seen in the first 48 hours after the second vaccination (11). In contrast, in a prospective study from Germany with the same vaccination strategy, they identified a comparable reactogenicity between heterologous (Astra Zeneca vaccine/Pfizer vaccine) and homologous (Pfizer vaccine/Pfizer vaccine) booster vaccination after a 12-week dose interval (12). On the other hand, participants receive an overview of their own immune response after vaccination at several time points and their participation contributes to answering a very relevant research question. The burden of the study visits is expected to be minimal.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give written informed consent for participation in the trial.
2. Adult (male/female) between 18 and 65 years old
3. Sufficient level of the Dutch language to undertake all study requirements

Exclusion Criteria:

1. Adults younger than 18 or older than 65 years
2. Adults already vaccinated with other vaccine then Janssen
3. Previously had a COVID-19 infection
4. History of allergic reaction likely to be exacerbated by any component of study vaccines (e.g. hypersensitivity to the active substance or any of the ingredients of the Janssen/Pfizer/Moderna vaccine).
5. Adults that are pregnant or have a wish to become pregnant within 6 months
6. Currently being treated for cancer
7. Severe kidney failure or dialyses dependent
8. Status after organ-, stem cell- or bone marrow transplantation
9. Use of immunosuppressant's
10. Epilepsy
11. HIV
12. Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding of bruising following injections of vene puncture
13. Continuous use of anticoagulants, such as coumarins (e.g. acenocoumarol) or novel oral anticoagulants (i.e. apixaban, dabigatran etc).
14. Participants who are currently participating in another research trial.
15. All regular contra-indications of the vaccines will be applied.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Determination of antibodies by a quantitative IgG assay (LIAISON SARS-CoV-2 TrimericS IgG essay) 28 days after booster | 28 days after booster
  LIAISON® SARS-CoV-2 TrimericS IgG assay

CONTACTS AND LOCATIONS:
Overall Officials: Hugo van der Kuy, PhD, PharmD, Principal Investigator — Erasmus Medical Center
Locations (4):
- Netherlands (4):
  - AmsterdamUMC, Amsterdam
  - UMCG, Groningen
  - LUMC, Leiden
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request to the study coordinator data will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available within 12 months after the end of the study.
Access Criteria: Reasonable request

REFERENCES:
- [Derived] Sablerolles RSG, Rietdijk WJR, Goorhuis A, Postma DF, Visser LG, Geers D, Schmitz KS, Garcia Garrido HM, Koopmans MPG, Dalm VASH, Kootstra NA, Huckriede ALW, Lafeber M, van Baarle D, GeurtsvanKessel CH, de Vries RD, van der Kuy PHM; SWITCH Research Group. Immunogenicity and Reactogenicity of Vaccine Boosters after Ad26.COV2.S Priming. N Engl J Med. 2022 Mar 10;386(10):951-963. doi: 10.1056/NEJMoa2116747. Epub 2022 Jan 19. PMID 35045226